CLINICAL TRIAL: NCT03023735
Title: Trial of Strategies to Communicate Genetic Information to Different Ethnic and Racial Subpopulations
Brief Title: Trial of Strategies to Communicate Genetic Information to Different Ethnic Subpopulations
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Stanford University (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, VJ Periyakoil, Clinical Associate Professor, Stanford University
Other Study IDs: 37046
Record Dates: First submitted 2017-01-06; First posted 2017-01-18 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: None. This is an observational study

SUMMARY:
The goal of this study is to better understand how clinicians give genetic risk information to patients from multi-ethnic groups and how patients understand this information and remember it and act upon it. In addition investigators want to know how to better communicate with patients about complex health issues across the health literacy divide and communication gap that exists between doctors and their patients.

DETAILED DESCRIPTION:
Any patient referred to the breast cancer and genetic risk counseling clinics in either of the two sites will be eligible to participate as long as they meet the inclusion and exclusion criteria. The research assistant in each site will meet with the patients and explain about the study goals and procedures and ask them to participate in the study. Those interested will be enrolled into the study after obtaining informed consent. For those who refuse to participate, reasons for refusal will be requested and catalogued. All study participants will be followed and the study measures will be tracked at Days 0, 30, 180 and 365. In addition, health care utilization (ER Visits, Hospitalizations, clinic visits, screening tests and procedures) will be tracked both through the electronic medical records and patient interviews (as some patients may seek care in other hospitals for emergencies etc.). Investigators currently do follow-up phone interviews routinely with our patients. Study measures will be administered as described above. For those who drop out from the study, reasons for withdrawal from the study will be explored and catalogued.

Procedures for Treatment Compliance and Treatment Non-completers:

(i) Compliance Procedures: Investigators will monitor degree of compliance with whether study measures were completed on Days 0,7,30 & 365 intervention. Analyses will be done following the intent-to-treat principle.

(ii) Treatment Non-completers: For those who drop out from the study after Day 0, reasons for withdrawal from the study will be explored and catalogued. They will be asked for feedback about the study intervention and satisfaction with the experience (or the lack thereof).

Procedures for Data Collection: The participants will have the option of submitting the data in person or by phone to the project research associate. The PI will meet with the study personnel at least on a weekly basis to continuously monitor their performance and to ensure adherence to study methodology.

There are risks, discomforts, and inconveniences associated with any research study. These deserve careful thought. Participants should talk with the Protocol Director for any questions. Risks of answering the survey instruments and interview questions are minimal and may occasionally cause distress.

Audio recording of the patient interviews. Investigators will create verbatim transcripts to be analyzed using qualitative methods. Recordings will be stored for a period of 20 years and then erased.

ELIGIBILITY:
Inclusion Criteria:

* Cancer Patients
* Over 18 years of age.

Exclusion Criteria:

* Under 18
* Healthy Volunteers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient referred to the breast cancer genetic risk counseling clinics in either of the two sites will be eligible to participate as long as they meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2016-08; Primary Completion 2023-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Composite outcome measure using health decisions and healthcare utilization | up to 3 years
  In this observational study, investigators propose to follow patients for a period of one to three years to track their cancer treatment and screening decisions (e.g. if they complete mammograms, MRI, surgery, chemotherapy, radiation therapy) as recommended by the clinical team and also ER visits, hospitalizations, ICU admissions and death.

CONTACTS AND LOCATIONS:
Overall Officials: VJ Periyakoil, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided